CLINICAL TRIAL: NCT04354012
Title: Prospective Case Series on a Combination Methylene Blue, Gentian Violet, and Ovine Forestomach-derived Extracellular Matrix Dressing for Hidradenitis Suppurativa
Brief Title: Hidradenitis Suppurativa Wound Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00063673
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-08

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Methylene Blue; Gentian Violet

STUDY DESIGN:
Intervention Model Description: Case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): methylene blue, gentian violet, and ovine forestomach wound dressings to HS lesions
  Interventions: Combination Product: methylene blue, gentian violet, and ovine forestomach wound dressings

INTERVENTIONS:
Combination Product: methylene blue, gentian violet, and ovine forestomach wound dressings — Hydrofera Blue is an antibacterial foam dressing that contains methylene blue and gentian violet to manage wounds. This is a safe, non-cytotoxic product that can be worn for 7 days while not inhibiting growth factors. This products wicks bacteria into the foam and away from the wound surface using natural negative pressure through capillary flow.
  Endoform (ovine forestomach) is a natural dermal template used in all phases of wound healing. This product helps to stabilize, build, and organize tissue in acute and chronic wounds.
  Hypafix tape aids in stabilization of wound dressings. This productIt is easy to apply, skin friendly, and comfortable to use.

SUMMARY:
The objective of this case series is to monitor time and outcome of healing of wounds associated with HS using Endoform [ovine forestomach], Hydrofera Blue [methylene blue and gentian violet], and Hypafix tape. a combination methylene blue, gentian violet, and ovine forestomach wound care product.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic and debilitating inflammatory disease most frequently affecting the axilla, groin, and inframammary regions. Symptoms include nodules, abscesses, sinus tract formation, malodorous drainage, and scarring. These symptoms interfere with everyday activities, which can lead to social embarrassment and isolation. Patients with HS suffer psychological effects, such as increased levels of anxiety, depression, and loneliness, which impair quality of life.

Patients suffer with the burden of at home wound care for recurrent, draining nodules. Persistent lesions affect patients' lives by limiting their daily activities. Currently, patients are instructed to use gauze and tape to cover draining wounds, but this can be insufficient and difficult due to the nature and location of lesions associated with HS. Patients suffer with caring for their wounds, which can lead to frustration. Providing patients with a standard wound care regimen to take home can improve patients' quality of life and control of their disease. General recommendations for wound care in HS patients are limited. Improvements in the standard of care for wound management in HS are needed to aid patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with hidradenitis suppurativa with non-healing wounds or draining abscesses/nodules
* Individuals over 18 years of age

Exclusion Criteria:

* Individuals younger than 18 years of age
* Individuals without a diagnosis of HS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita O Pichardo, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study to determine use and outcomes; the plan is to be able to provide overall group data since it is such a small set of participants.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: methylene blue, gentian violet, and ovine forestomach wound dressings to HS lesions
  methylene blue, gentian violet, and ovine forestomach wound dressings: Hydrofera Blue is an antibacterial foam dressing that contains methylene blue and gentian violet to manage wounds. This is a safe, non-cytotoxic product that can be worn for 7 days while not inhibiting growth factors. This products wicks bacteria into the foam and away from the wound surface using natural negative pressure through capillary flow.
  Endoform (ovine forestomach) is a natural dermal template used in all phases of wound healing. This product helps to stabilize, build, and organize tissue in acute and chronic wounds.
  Hypafix tape aids in stabilization of wound dressings. This productIt is easy to apply, skin friendly, and comfortable to use.
Period: Overall Study
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 37.8 [19 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Wound Size
Description: Asses the percent healing that occurs over 8 weeks of follow-up using Endoform and Hydrofera Blue products
Time Frame: Measure from Baseline to week 8
Measure: Mean (Full Range); unit: percentage change in wound size
Arm/Group | Treatment
Number analyzed (Participants) | 5
percentage change in wound size | 57.2 [4.6 to 100]

2. Secondary Outcome: Change in Pain Assessment Scores
Description: Assess changes in patient reported pain via Numerical Rating Scale of Pain (NRS) a scale using a number from 0 to 10 where 0 is no pain or hurt and 10 is the most or worst pain.
Time Frame: Change from baseline to week 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 5
score on a scale | 5 [0 to 8]

3. Secondary Outcome: Change in Pain Assessment Scores
Description: as for outcome 2
Time Frame: Change from week1 to week 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 5
score on a scale | 3.8 [0 to 8]

4. Secondary Outcome: Change in Pain Assessment Scores
Description: as for outcome 2
Time Frame: Change from week 2 to week 4
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 5
score on a scale | 4.2 [0 to 8]

5. Secondary Outcome: Change in Pain Assessment Scores
Description: as for outcome 2
Time Frame: Change from week 4 to week 8
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 4
score on a scale | 3.12 [0 to 8]

6. Post Hoc Outcome: Wound Healing Time
Description: Assess the time for wound healing to occur using Endoform and Hydrofera Blue products.
Time Frame: Change from week 4 to week 8
Population: Wound Healing Time was not analyzed
Arm/Group | Treatment
Number analyzed (Participants) | 0

7. Post Hoc Outcome: Wound Healing Time
Description: Assess the time for wound healing to occur using Endoform and Hydrofera Blue products.
Time Frame: Change from week 2 to week 4
Population: Wound Healing Time was not analyzed
Arm/Group | Treatment
Number analyzed (Participants) | 0

8. Post Hoc Outcome: Wound Healing Time
Description: Assess the time for wound healing to occur using Endoform and Hydrofera Blue products.
Time Frame: Change from week 1 to week 2
Population: Wound Healing Time was not analyzed
Arm/Group | Treatment
Number analyzed (Participants) | 0

9. Post Hoc Outcome: Wound Healing Time
Description: Assess the time for wound healing to occur using Endoform and Hydrofera Blue products.
Time Frame: Change from baseline to week 1
Population: Wound Healing Time was not analyzed
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline, 1 week, 2 week, 4 week, 8 week
Description: There were no adverse events report
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT04354012/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT04354012/ICF_000.pdf